CLINICAL TRIAL: NCT07234279
Title: Feasibility of the Investigational Nellcor™ Investigational Device During Non-Motion and Walking Motion Conditions in Adult Volunteers
Brief Title: Nellcor™ Investigational Device Sitting-Walking Study
Status: Not yet recruiting | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT25003NPDSWF
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Oxygen Saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy Volunteers: All subjects who meet the inclusion criteria and none of the exclusion criteria will be enrolled into the test group and will participate in data collection with use of the Nellcor™ Investigational device.

SUMMARY:
To examine pulse rate and blood oxygen saturation accuracy of the Nellcor™ Investigational Device during non-motion and walking motion conditions in a diverse patient population through non-invasive means

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥18 years of age, and <75 years of age.
* Participant is able to participate for the duration of the study
* Participant is willing to sign an informed consent form (ICF)
* Participant weighs > 40kg
* Participants must be a non-smoker or not have smoked within 36 hours prior to the study

Exclusion Criteria:

* Participant self-reported prior injury or trauma to fingers or hands, which in the opinion of the investigator, may change blood flow or vascular supply and affect the ability to test sensors
* Physiologic abnormalities that prevent proper application of pulse oximetry sensor
* Severe contact allergies that cause a reaction to standard adhesive materials such as those found in medical sensors and electrodes
* Individuals of childbearing potential who are self-reported as pregnant, or who are self-reported as trying to get pregnant
* Morbid obesity (defined as BMI > 39.5)
* Weight > 136 kg
* Participants who self-report problems of unsteadiness or imbalance issues and/or who are unable to walk on a treadmill without holding onto the handrails
* Participant self-reported known heart or cardiovascular conditions such as:
* Uncontrolled hypertension (Systolic pressure ≥ 140mmHg or Diastolic pressure > 90mmHg on 3 consecutive readings day of screening)
* Heart arrhythmias other than sinus arrhythmia (Self-reported and/or as identified on ECG day of screening).
* History of heart attack, blocked artery, history of myocardial ischemia, angina, myocardial infarction, congestive heart failure, cardiomyopathy, stroke, transient ischemic attack, or carotid artery disease
* Participants with self-reported clotting disorders, such as:
* History of bleeding disorders or personal history of prolonged bleeding from injury
* History of blood clots
* Hemophilia
* Current use of prescription blood thinner
* Participants with other self-reported, known health conditions, such as:
* Diabetes
* Thyroid disease
* Kidney disease / chronic renal impairment
* History of seizures (except childhood febrile seizures), epilepsy, or unexplained syncope
* Recent history of frequent migraine headaches, as determined medically relevant by the PI
* History of head injury, as determined medically relevant by the PI
* Cancer / chemotherapy
* Sickle cell disease
* History of hospital admission or a surgical procedure in the 60 days prior to study enrollment (self-reported)
* Participants with any contraindications to protocol specific repositioning techniques
* Unwillingness or inability to remove colored nail polish from test digit(s)
* Participants who have self-reported health conditions beyond what is captured in the prior exclusion criteria, which in the opinion of the Investigator and/or Clinical Staff would classify the participant as medically unsuitable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the investigational device SpO2 as compared to the reference device SpO2 | From enrollment to study exit, 1.5 hours
Accuracy of the investigational device pulse rate as compared to the reference device pulse rate. | From enrollment to study exit, 1.5 hours

SECONDARY OUTCOMES:
Percentage of the time under evaluation that the NellcorTM Investigational Device provides a SpO2 and PR reading | From enrollment to study exit, 1.5 hours

IPD SHARING:
Plan to Share IPD: No